CLINICAL TRIAL: NCT05592535
Title: Prognostic Impact of Fractional Flow Reserve in Chronic Coronary Syndrome: Quasi-Experimental Findings Using a Regression Discontinuity Design
Brief Title: Outcomes With Fractional Flow Reserve in Chronic Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2022-10-17; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Chronic Coronary Syndrome
Keywords: Percutaneous Coronary Intervention; Fractional Flow Reserve
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FFR below 0.80: Patients with significant coronary hyperemic gradient
  Interventions: Procedure: Coronary revascularization
- FFR above 0.80: Patients without significant coronary hyperemic gradient

INTERVENTIONS:
Procedure: Coronary revascularization — Coronary revascularization performed by PCI in a vessel investigated with FFR or indication for surgery
  Groups: FFR below 0.80

SUMMARY:
The use of fractional flow reserve (FFR) to assess the functional relevance of coronary stenoses has been demonstrated to reduce the risk urgent revascularization in chronic coronary syndrome patients.[1] The goal of this study is to assess whether the utility of using FFR during percutaneous coronary intervention (PCI) in chronic coronary syndrome patients is confirmed in a real-life scenario. This study will implement a regression discontinuity design (RDD). RDD is a quasi-experimental study design able to provide robust findings on causality using observational data.

DETAILED DESCRIPTION:
All patients in this study were included in the Swedish Coronary Angiography and Angioplasty Registry (SCAAR), a sub-registry of SWEDEHEART. [2] Data regarding FFR assessments are documented in SCAAR in terms of FFR values and coronary segments investigated with FFR. The use of FFR during PCI is left at the discretion of the operator. Since a nondeterministic assignment to revascularization is expected at the cut-off, a fuzzy RDD design will be used in the analyses. Moreover, FFR values equal to 0.80 (at the cut-off) will be excluded from the analysis since treatment assignment exactly at the cut-off may substantially vary across operators and this may create distortions in the treatment discontinuity. Local linear regression estimates with Kernel triangulation and asymmetric bandwidth selection will be used in the analysis. Bandwidth selection will be based on a fully data-driven approach that minimizes the bias-variance trade-off.[3] Estimates from RDD will be presented as risk differences [RD] complemented by 95% robust confidence intervals.[4]

ELIGIBILITY:
Inclusion Criteria:

* Chronic coronary syndrome undergoing coronary angiography and FFR measurement
* Swedish personal identification number

Exclusion Criteria:

* previous coronary artery bypass grafting
* left main disease or undergoing FFR/PCI of left main
* IVUS/OCT use
* diffuse disease (≥ 2 segments treated in a same vessel investigated with FFR, ≥ 2 segments investigated with FFR in a same vessel)
* PCI in a distal segment with respect to FFR measurements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic coronary syndrome undergoing coronary angiography and FFR measurement in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Risk difference (%) for the composite of all-cause death and FFR-oriented target vessel revascularization by PCI | Up to one year following index FFR measurement

SECONDARY OUTCOMES:
Risk difference (%) for the composite of all-cause death, FFR-oriented target vessel revascularization by PCI and hospitalization for acute myocardial infarction | Up to one year following index FFR measurement
Risk difference (%) for the composite of all-cause death and new hospitalization for acute myocardial infarction | Up to one year following index FFR measurement
Risk differences (%) for the individual components of the composite outcome measures | Up to one year following index FFR measurement

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638
- [Background] Jernberg T, Attebring MF, Hambraeus K, Ivert T, James S, Jeppsson A, Lagerqvist B, Lindahl B, Stenestrand U, Wallentin L. The Swedish Web-system for enhancement and development of evidence-based care in heart disease evaluated according to recommended therapies (SWEDEHEART). Heart. 2010 Oct;96(20):1617-21. doi: 10.1136/hrt.2010.198804. Epub 2010 Aug 27. PMID 20801780
- [Background] Calonico S, Cattaneo MD, Farrell MH. Optimal bandwidth choice for robust bias corrected inference in regression discontinuity designs. Econom J. 2020;23(2):192-210.
- [Background] Calonico S, Cattaneo MD, Titiunik R. Robust nonparametric confidence intervals for regression-discontinuity designs. Econometrica. 2014;82(6):2295-2326.